CLINICAL TRIAL: NCT07191028
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parellel-group Study to Assess the Efficacy and Safety of MLC901 (NeuroAiD™II) in Subjects With Mild to Moderate Alzheimer's Disease (AD).
Brief Title: Alzheimer's Disease THErapy With NEuroaid II
Acronym: ATHENE II
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Moleac Pte Ltd. (Industry)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFSA2025_01
Record Dates: First submitted 2025-09-02; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease Dementia
Keywords: MLC901; NeuroAiD™II; Alzheimer's disease; multicenter; randomised; double blind; placebo controlled
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuroaid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parellel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study partner and sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MLC901 (Experimental): Active arm
  Interventions: Drug: MLC 901
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MLC 901 — Oral capsule, 2 capsules 3 times a day for 12 months
  Arms: MLC901
Drug: Placebo — Oral capsule, 2 capsules 3 times a day for 12 months
  Arms: Placebo

SUMMARY:
ATHENE II is a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial designed to evaluate the efficacy and safety of MLC901 in subjects with mild to moderate Alzheimer's disease, as well as its effects on plasma biomarkers compared to placebo.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive neurodegenerative disorder with limited treatments that slow progression. Current symptomatic therapies provide modest benefit, while anti-amyloid agents target a single pathway and have uncertain long-term outcomes. Multitarget approaches may provide broader and more durable benefit. MLC901 (NeuroAiD™II), a Traditional Chinese Medicine derived formulation, has shown neuroprotective and neuroproliferative properties in preclinical studies through multimodal mechanisms, including modulation of amyloid beta and tau phosphorylation, reduction of oxidative stress and inflammation, and promotion of neurogenesis and synaptogenesis. Clinical studies, including the ATHENE trial, suggest MLC901 may slow cognitive decline and is well tolerated. ATHENE II is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study enrolling approximately 350 patients with mild to moderate AD across Southeast Asia. Participants will receive MLC901 or placebo for 12 months. The primary objective is to determine whether MLC901 is superior to placebo in slowing cognitive decline as measured by ADAS-Cog14. Secondary and exploratory objectives include global cognition, function, behavior, safety, and plasma biomarkers of AD (p-tau217, NfL and GFAP).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 50 years at the time of providing informed consent.
* Diagnosis of AD based on the National Institute on Ageing and the Alzheimer's Association criteria, supported by the presence of a Core 1 AD biomarker, specifically elevated plasma ptau217.
* MMSE score between 10 and 26, inclusive, at baseline, corresponding to mild to moderate AD.
* Subjects may be either treatment-naïve or currently receiving stable symptomatic treatment for AD for at least the 2 months prior to screening, including AChEIs, memantine, or a combination of both.
* Subjects must have a designated study partner who provides ongoing support during the study and interacts with the subject for a minimum of 8 hours per week, and will accompany the subject to study visits or be available by telephone at designated times. A second study partner may serve as backup. If the original study partner withdraws from participation, a replacement study partner may be permitted at the investigator's discretion. The replacement study partner must provide informed consent prior to their first study visit with the subject.
* Both the subject (or their legally authorized representative) and the study partner(s) must be capable of providing informed consent.
* Subjects must have adequate literacy, vision, and hearing, in the opinion of the investigator at the time of screening, to allow for valid administration of the clinical outcome assessments.

Exclusion Criteria:

* Presence of any neurological disorder contributing to cognitive impairment other than AD, including but not limited to: Parkinson's disease, Dementia with Lewy bodies, and epilepsy or recurrent seizures.
* Evidence of other clinically significant cerebrovascular disease or intracranial abnormalities based on the latest brain CT or MRI, including but not limited to: multiple lacunar infarcts, large territorial infarcts, severe small vessel or white matter disease, normal pressure hydrocephalus, space occupying lesions.

The most recent available scan (obtained at diagnosis or subsequently) is usually sufficient for screening eligibility to exclude these other conditions. Repeat imaging may need in some cases to be considered if there is clinically significant deterioration or new neurological signs suggestive of a cerebrovascular event.

* Presence of any serious or unstable medical illnesses, including but not limited to: cardiovascular, respiratory, gastroenterological, endocrinologic, immunologic, hematologic, hepatic, or renal and other conditions, that, in the investigator's judgment, may interfere with study participation or compromise subject safety.
* Patients with a CDR Global Score of 0, 0.5 or 3 at the Screening Phase, corresponding to no, very mild or severe dementia, respectively, will be excluded from the study.
* Severe visual or hearing impairment that would prevent the subject from accurately completing clinical outcome assessments.
* Serum creatinine > 130 µmol/L at baseline, which may affect plasma biomarker analysis.
* Female subjects who are pregnant at screening.
* Participation in another clinical trial or receipt of any investigational product within 60 days or 5 half-lives (whichever is longer) prior to screening.
* Current use at baseline of any AD disease-modifying therapies or neuroprotective/nootropic agents, including Ginkgo biloba, Neurotain, Citicoline, Cerebrolysin, or Piracetam.
* Known hypersensitivity or allergic reaction to MLC901 or any of its components. Any known food allergy or hypersensitivity to Astragalus membranaceus, Ligusticum chuanxiong, Polygala tenuifolia, Angelica sinensis or members of the Fabaceae/Leguminosae family (e.g., legume, pea, bean), Polygalaceae family (e.g., milkwort, snakeroot), Apiaceae/Umbelliferae family (e.g., anise, caraway, carrot, celery, dill, parsley, parsnip) or Quillaja bark (soapbark).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive Subscale14 (ADAS-Cog14) | Baseline, Month 3, Month 6, Month 9 and Month 12
  The ADAS-Cog is a rater-administered instrument designed to assess the severity of cognitive impairment and associated non-cognitive behaviors characteristic of individuals with AD. It is the most widely used cognitive scale in clinical trials evaluating treatments for mild to moderate AD.
  For this study, the version of ADAS-Cog14 will be used as the primary efficacy assessment. The ADAS-Cog14 consists of 14 items assessing key areas of cognitive function that are commonly impaired in AD, including: orientation, word recall, word recognition, remembering word recognition test instructions, commands, comprehension of spoken language, naming, word-finding difficulty, spoken language ability, construction praxis, ideational praxis, delayed word recall, number cancellation and maze completion measures.
  The ADAS-Cog14 total score ranges from 0 to 90, with higher scores indicating greater cognitive impairment.

SECONDARY OUTCOMES:
Clinical Dementia Rating (CDR): Global Score and Sum of Boxes (CDR-SB) | Baseline, Month 6 and Month 12
  The CDR evaluates both cognitive and functional domains through structured interviews conducted with both the participant and a knowledgeable informant (such as a caregiver or study partner). The assessment is administered by a trained assessor according to a standardized protocol. The CDR includes the following 6 domains: 3 cognitive domains (memory, orientation, and judgment/problem solving) and 3 functional domains (community activities, home and leisure, and personal care). Each domain is rated on a scale from 0 (no impairment) to 3 (severe impairment). The CDR yield 2 scores, including CDR Global Score and CDR-SB. The CDR global score: a categorical rating from 0 to 3, derived via a standardized algorithm. This score is used to stage the severity of dementia as follows: 0= No dementia; 0.5= Very mild dementia; 1= Mild dementia; 2= Moderate dementia; 3= Severe dementia. CDR-SB: a continuous score ranging from 0 to 18, calculated by summing the individual domain scores.
Mini-Mental State Examination (MMSE) | Baseline, Month 3, Month 6, Month 9 and Month 12
  The MMSE, developed by Folstein et al. in 1975, is a brief and widely used tool for evaluating global cognitive function. The MMSE assesses multiple cognitive domains, including orientation, memory, attention, object naming, the ability to follow verbal and written instructions, sentence writing, and figure copying. The total MMSE score ranges from 0 to 30, with lower scores indicating greater cognitive impairment.
Montreal Cognitive Assessment (MoCA) | Baseline, Month 3, Month 6, Month 9 and Month 12
  The MoCA test was validated as a highly sensitive tool for the early detection of MCI. It is widely used in both clinical and research settings to assess global cognitive function. The MoCA evaluates the following cognitive domains: short-term memory, visuospatial abilities, executive functions, language, orientation to time and place and attention, concentration and working memory. The total MoCA score ranges from 0 to 30, with lower scores indicating greater cognitive impairment.
Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Baseline, Month 6 and Month 12
  The ADCS-ADL, developed by Galasko et al, is the most widely used instrument for assessing functional outcomes in patients with AD. This 23-item scale evaluates both basic activities of daily living-such as eating and toileting-and more complex instrumental activities of daily living. The ADCS-ADL is administered as a structured interview with the participant's study partner or caregiver. For each item, the study partner is first asked whether the participant attempted the activity within the past four weeks. If so, the study partner is then asked to describe the participant's performance, which is scored accordingly.
  The total ADCS-ADL score ranges from 0 to 78, with lower scores indicating greater functional impairment.
Neuropsychiatric Inventory (NPI) | Baseline, Month 6 and Month 12
  The NPI is a validated instrument developed to assess a broad spectrum of behavioral and psychological symptoms commonly observed in individuals with dementia. The purpose of the NPI is to characterize the presence and severity of these symptoms. The questionnaire assesses 12 neuropsychiatric symptom domains: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, aberrant motor behavior, nighttime disturbances, and appetite/eating abnormalities.
  For each symptom domain, both frequency and severity are assessed. Severity is rated on a 3-point scale (mild, moderate, or marked), while caregiver distress related to each symptom is also rated on a 6-point scale (ranging from no distress to very severe distress). The NPI is administered via a structured interview with the subject's study partner or caregiver, who provides observations based on the subject's behavior.
Adverse events | Up to 52 weeks
  Listing and calculating the number and percentage of subjects experiencing non-serious and serious adverse events for each arm.

OTHER OUTCOMES:
Plasma biomarkers - phosphorylated tau (p-tau217) | Baseline, Month 6 and Month 12
  Plasma samples will be collected from all subjects and used for research purposes to identify dynamic biomarkers that may be predictive of treatment response to MLC901.
  During screening, at baseline and subsequent visits as detailed in the Schedule of Events, whole blood samples will be obtained from every subject who has consented to participate in the study. The plasma samples will be used to evaluate p-tau217 in pg/mL.
Plasma biomarkers - neurofilament light chain (NfL) | Baseline, Month 6 and Month 12
  Plasma samples will be collected from all subjects and used for research purposes to identify dynamic biomarkers that may be predictive of treatment response to MLC901.
  During screening, at baseline and subsequent visits as detailed in the Schedule of Events, whole blood samples will be obtained from every subject who has consented to participate in the study. The plasma samples will be used to evaluate NfL in pg/mL.
Plasma biomarkers - glial fibrillary acidic protein (GFAP) | Baseline, Month 6 and Month 12
  Plasma samples will be collected from all subjects and used for research purposes to identify dynamic biomarkers that may be predictive of treatment response to MLC901.
  During screening, at baseline and subsequent visits as detailed in the Schedule of Events, whole blood samples will be obtained from every subject who has consented to participate in the study. The plasma samples will be used to evaluate GFAP in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Li Hsian Chen, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) for this study. Only de-identified, aggregate study findings will be disseminated through scientific meetings and peer-reviewed publications.

REFERENCES:
- [Background] Dib M, Ampil E, Kee HF, et al. A review of NeuroAiD™ II (MLC901) development in Alzheimer's disease treatment: promises of a multimodal pathway. J Neurol Res Rev Rep. 2022 Jun 30;1-13.
- [Background] Lee WT, Hsian CCL, Lim YA. The effects of MLC901 on tau phosphorylation. Neuroreport. 2017 Nov 8;28(16):1043-1048. doi: 10.1097/WNR.0000000000000884. PMID 28902708
- [Background] Lim YA, Murray LA, Lai MK, Chen C. NeuroAiD(R) (MLC601) and amyloid precursor protein processing. Cerebrovasc Dis. 2013;35 Suppl 1:30-7. doi: 10.1159/000346236. Epub 2013 Mar 14. PMID 23548917
- [Background] Heurteaux C, Widmann C, Moha ou Maati H, Quintard H, Gandin C, Borsotto M, Veyssiere J, Onteniente B, Lazdunski M. NeuroAiD: properties for neuroprotection and neurorepair. Cerebrovasc Dis. 2013;35 Suppl 1:1-7. doi: 10.1159/000346228. Epub 2013 Mar 14. PMID 23548913
- [Background] Heurteaux C, Gandin C, Borsotto M, Widmann C, Brau F, Lhuillier M, Onteniente B, Lazdunski M. Neuroprotective and neuroproliferative activities of NeuroAid (MLC601, MLC901), a Chinese medicine, in vitro and in vivo. Neuropharmacology. 2010 Jun;58(7):987-1001. doi: 10.1016/j.neuropharm.2010.01.001. Epub 2010 Jan 11. PMID 20064536